CLINICAL TRIAL: NCT05832801
Title: Effect of Pilates Exercises on Symptom Severity in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Pilates Exercises on Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Mohammed Mahmoud Allam, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004218
Record Dates: First submitted 2023-03-29; First posted 2023-04-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into two groups, group A and group B .Patients in both groups will receive a traditional dietary advice for IBS, but group (A) will receive additional pilates exercises.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ( Traditional dietary advice) (Other): Each patient will follow traditional dietary advice only for 2 months.
  Interventions: Other: ( Traditional dietary advice )
- Group (Pilates and traditional dietary advice ) (Experimental): Patients in this group will participate in 2 months Pilates exercise program, 2 times per week for 16 sessions, and will follow traditional dietary advice. Warming up and cooling down stretches for 5 minutes will be done before and after exercise .
  Interventions: Other: ( Traditional dietary advice ); Other: (Pilates exercises)

INTERVENTIONS:
Other: ( Traditional dietary advice ) — traditional dietary advice for IBS which is based on guidance provided by the National Institute for Health and Care Excellence (NICE ) and the British Dietetic Association (BDA). Its principles include adopting healthy, sensible eating patterns such as having regular meals, never eating too little/too much, maintaining adequate hydration, and reducing the intake of (1) alcohol/caffeine/fizzy drinks, (2) fatty/spicy/processed foods, (3) fresh fruit to a maximum of 3 per day, (4) fiber and other commonly consumed gas-producing foods (eg, beans, bread, sweeteners, etc), and (5) addressing any perceived food intolerances (eg, dairy).
Other: (Pilates exercises) — Pilates exercises will be in the form of Swan, One leg up-down, Leg circles, Single leg stretch, Saw, Side kicks, The hundred,. Pelvic lift on the ball, Sit-ups with the ball, Stretching on the ball. exercise Dose will be First month (first- eighth session) composed of one set of eight repetitions Second month (eighth-sixteenth session) composed of two sets of ten repetitions
  Arms: Group (Pilates and traditional dietary advice )

SUMMARY:
purpose: to investigate the effect of pilates exercises on patients with irritable bowel syndrome. Methods sixty patients with IBS will be recruited and randomly assigned into two groups, group A and group B. Patients in both groups will receive a traditional dietary advice for IBS, but group A will receive additional pilates exercises. All patients will be evaluated pre and post treatment for irritable bowel syndrome symptom severity, number of bowel movements , anxiety and depression , Fatigue and body weight.

DETAILED DESCRIPTION:
A) Procedures for evaluation:

The practical section of the study will be undertaken in 2months (2 sessions a week). Measurement will be taken before the start of treatment program then after the end of 2 months of treatment program in the following manner:

1. -Irritable bowel syndrome symptom severity score (IBS-SSS) will be used to measure severity of IBS symptoms
2. number of bowel movements per week will be recorded
3. The hospital anxiety and depression scale will be used to assess depression and anxiety
4. Modified Fatigue Impact scale (MFIS): was developed to assess the perceived impact of fatigue on a variety of daily activities.
5. weight height scale for assessing BMI

B-Treatment procedures:

All patients in both groups will be instructed to follow traditional dietary advice for IBS which is based on guidance provided by the National Institute for Health and Care Excellence (NICE ) and the British Dietetic Association (BDA). .

Group (A) Patients in this group will participate in 2 months Pilates exercise program, 2 times per week for 16 sessions, and will follow traditional dietary advice for IBS. Warming up and cooling down stretches for 5 minutes will be done before and after exercise Group (B) Each patient will follow traditional dietary advice for IBS which is based on guidance provided by the National Institute for Health and Care Excellence (NICE ) and the British Dietetic Association (BDA).

C)Data analysis: Statistical analysis will be performed through the statistical package for social studies (SPSS) version 24 for windows. Descriptive statistics will be conducted to describe the data. Mixed-Model ANOVA will be used to determine the within-group changes and the between-group difference. The level of significance for all statistical tests will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. They will be under medical supervision.
2. Age between 20 to 45 years.).
3. Ability to perform exercises.
4. Diagnosis of IBS will be based on Rome IV Diagnostic criteria.
5. Baseline irritable bowel syndrome severity score >174
6. over weight or grade one obese IBS patients who diagnosed as constipation predominant IBS according to Bristol stool scale.

Exclusion Criteria:

1. Organic gastrointestinal disorders or other organic disease hindering physical activity.
2. Treatment with steroids, immunosuppressants for at least 6 months before the beginning of the study.
3. A history of resection of the stomach, small intestine, or large intestine .
4. Concurrent infectious enteritis, hyperthyroidism, hypothyroidism, or other diseases that may affect gastrointestinal transit or colonic function.
5. History or current evidence of abuse of drugs or alcohol within the previous year.
6. Malignant tumors.
7. Concurrent serious cardiovascular, respiratory, renal, hepatic, gastrointestinal (excluding IBS).
8. Fibromyalgia and pregnancy -

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Irritable bowel syndrome symptom severity | (at baseline and after 8 weeks)
  BS-SSS is a patient-based scale that assesses 5 clinically relevant items during a 10-day period: (1) severity of abdominal pain, (2) frequency of abdominal pain, (3) severity of abdominal distention or tightness, (4) dissatisfaction with bowel habits, and (5) interference of IBS with life in general. Each item is scored on a visual analogue scale (VAS) from 0 to 100, yielding overall scores ranging from 0 to 500 (a higher score indicates worse condition). A reduction of 50 in the IBS-score is adequate to detect a clinical improvement

SECONDARY OUTCOMES:
number of Bowel movement | (at baseline and after 8 weeks)
  Bristol stool form scale will be used to record bowel movements. The patients will record all bowel movements and its consistency The scale ranges from 1 to 7, where type 1 and 2 is hard and lumpy stools and type 6 and 7 is loose and watery stools
Anxiety and depression | (at baseline and after 8 weeks)
  Hospital Anxiety and Depression Scale(HADS), the HADS includes 14 items assessing anxiety (7-item) and depression (7-item), which are rated on a 4-point Likert-type (from 0 to 3).A score of 0-7 is considered as normal, 8-10 as a borderline case, and 11-21 as a case (anxiety or depression)
Fatigue | (at baseline and after 8 weeks)
  modified Fatigue Impact Scale, a multidimensional scale developed to assess the perceived impact of fatigue on a variety of daily activities. These scores are designed to measure the disability associated with fatigue (the extent to which fatigue limits activities), not the severity of symptoms. MFIS total score ranges from 0 to 20, with the following ranges reflecting how often the person is limited in activities by fatigue: 0 -5 (never), 6 -9 (rarely), 10-14 (sometimes), 15-19 (often) and 20 (almost always).
body weight | (at baseline and after 8 weeks)
  weight height scale used to assess body weight

CONTACTS AND LOCATIONS:
Overall Officials: Heba A. Abd El Ghafar, A. Professor, Study Director — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No